CLINICAL TRIAL: NCT03117439
Title: (1-3)-Beta-D-Glucan Driven vs. Empirical Antifungal Therapy in High Risk Critically Ill Patients A Randomized Study
Brief Title: Beta-Glucan Driven vs. Empirical Antifungal Therapy in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 100452
Record Dates: First submitted 2017-04-12; First posted 2017-04-18 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Antifungal Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Patients undergoing empirical anti fungal therapy. Interruption of anti fungal treatment will be decided on the basis of standard clinically and microbiologically criteria.
- 1-3 Beta-D-Glucan Group (Experimental): Patients undergoing anti fungal de-escalation according to 1-3 Beta-D-Glucan results
  Interventions: Other: duration of antifungal therapy

INTERVENTIONS:
Other: duration of antifungal therapy — Patients in the study group will stop antifungals in presence of a negative result of Beta Glucan Test
  Arms: 1-3 Beta-D-Glucan Group

SUMMARY:
This study is aimed to compare the duration of standard anti fungal therapy in high risk ICU patients with a strategy driven by BetaDGlucan test result

ELIGIBILITY:
Inclusion Criteria:

* ICU admission (minimum of 48 hours in ICU with an expected length of stay of at least 48 hours)
* Ongoing Mechanical Ventilation
* Presence of CVC
* Sepsis/Septic Shock development while receiving broad spectrum antibiotics
* Positivity of Candida Score or Candida Colonization Index in absence of septic shock

Exclusion Criteria:

* Complicated Candida Infection
* Already ongoing anti fungal therapy
* Beta Glucan test not available
* Absence of informed consent
* Immunesuppressive status (long-term immunesuppresive or steroids therapy; AIDS; WBC <1000/mmc or neutrophils <500/mmc)
* Pregnancy
* Already enrolled in other interventional studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Reduction of anti fungal duration in the Beta Glucan group compared with standard empirical approach | First 30 days from enrollment

SECONDARY OUTCOMES:
Clinical Cure of Invasive Canididiasis | 90 days
Microbiological eradication of Invasive Candidiasis | 90 days
30-day mortality | 30 days
ICU mortality | 90 days
  Any cause ICU mortality within three months from enrollment
Hospital mortality | 90 days
  Any cause hospital mortality within three months from enrollment
Duration of ICU length of stay | 90 days
Duration of mechanical ventilation | 90 days
Number of invasive Candida Infections and Beta-Glucan accuracy | 90 days
Cost evaluation (empirical anti fungal therapy vs. Beta Glucan test) | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Gennaro De Pascale, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Pascale G, Posteraro B, D'Arrigo S, Spinazzola G, Gaspari R, Bello G, Montini LM, Cutuli SL, Grieco DL, Di Gravio V, De Angelis G, Torelli R, De Carolis E, Tumbarello M, Sanguinetti M, Antonelli M. (1,3)-beta-D-Glucan-based empirical antifungal interruption in suspected invasive candidiasis: a randomized trial. Crit Care. 2020 Sep 5;24(1):550. doi: 10.1186/s13054-020-03265-y. PMID 32891170